CLINICAL TRIAL: NCT06827457
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Subcutaneous Injection of GenSci120 in Healthy Adult Participants in China
Brief Title: A Study of Safety, Tolerability, PK, and PD of Subcutaneous GenSci120 in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GenSci120-101
Record Dates: First submitted 2025-01-22; First posted 2025-02-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Disease
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GenSci120 (Experimental): Single ascending doses of GenSci120 administered subcutaneously (SC).
  Interventions: Drug: GenSci120
- Placebo (Placebo Comparator): Administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GenSci120 — Administered SC.
  Arms: GenSci120
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability, PK and PD of GenSci120 in a randomized, double-blind, placebo-controlled trial involving healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 55 years of age (inclusive) at the date of signed informed consent form (ICF), each cohort must include at least 3 participants of a single gender.
2. Body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and total body weight ≥ 50 kg (Male) / ≥ 45 kg (Female) at screening.
3. No clinically significant abnormalities in medical history, general physical examination, vital signs, laboratory tests (hematology, urinalysis, blood chemistry, coagulation function, tumor biomarker, et al.), electrocardiogram (ECG) and pulmonary imaging tests, or value beyond normal reference range considered not clinically significant.
4. Ability to understand the trial procedures, volunteer to participate in the trial, and could provide written informed consent.

Exclusion Criteria:

1. Known allergy to any component in the GenSci120 formulation, or a history of severe allergic reactions to any drugs, compounds, foods, or other substances, or a history of hypersensitivity.
2. The proposed injection site has tattoos, sunburn, scarring, or other factors that may interfere with the evaluation of the injection site.

(3) History of serious metabolic, allergic, dermatological, hepatic, renal, hematological, cardiovascular, gastrointestinal, neurological, respiratory, or other significant medical history that, in the investigator's opinion, may affect the assessment of this study.

（4）Severe infection, chronic infection, opportunistic infection, etc., within 3 months before screening, or systemic antimicrobial treatment for infections (including but not limited to viral, bacterial, fungal, parasitic infections) within 4 weeks prior to randomization.

（5）Use or intend to use any prescription medication to manage chronic/ongoing condition, and any acute medication use (including prescription medication, over-the-counter medication, or dietary supplements) within 14 days prior to administration.

（6)Participated in any clinical trials of investigational drugs (including investigational vaccines) and used investigational drugs within 3 months or within 5 terminal elimination half-lives (whichever is longer) prior to administration; participated in any clinical trials of medical devices within 3 months prior to screening (not including failed screening participants); currently participating in other clinical trials.

（7) Any other medical condition (at the investigator's discretion) that would impair the participant's ability to tolerate the IMP or proceed with the planned study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | 113 days
Incidence and severity of serious adverse events (SAEs) | 113 days
Clinically significant changes from baseline | 113 days
Concentration of GenSci120 in plasma samples. | 113 days
Pharmacokinetics-AUC0-last | 113 days
Pharmacokinetics-AUC0-inf | 113 days
Pharmacokinetics-Tmax | 113 days
Pharmacokinetics-Cmax | 113 days
Pharmacokinetics-CL/F | 113 days
Pharmacokinetics-t1/2 | 113 days
flow cytometry | 113 days
Incidence and the time of anti-drug antibody (ADA) positive and neutralizing antibody (NAb) positive (if applicable) after GenSci120 administration. | 113 days

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China